CLINICAL TRIAL: NCT00149045
Title: Clinical and Genetic Features of Familial Neuropathy
Brief Title: Follow up and Observation of Charcot Marie Tooth Disease in Families
Status: Completed | Type: Observational
Sponsor: Hadassah Medical Organization (Other)
Other Study IDs: 920010132-HMO-CTIL
Record Dates: First submitted 2005-09-07; First posted 2005-09-08 (Estimated); Last update posted 2006-11-07 (Estimated); Status verified 2005-08

CONDITIONS: Charcot-Marie-Tooth Disease
Keywords: familial peripheral Neuropathy Anticipation
MeSH Terms: conditions — Charcot-Marie-Tooth Disease

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
The study is aimed to test the hypothesis that there is anticipation in CMT

ELIGIBILITY:
Inclusion Criteria:Patients with Genetically confirmed CMT 1a disease -

Exclusion Criteria:

-

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2001-11; Study Completion 2005-08

CONTACTS AND LOCATIONS:
Overall Officials: Israel Steiner, MD, Principal Investigator — Hadssah University Hospital, Department of Neurology
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel